CLINICAL TRIAL: NCT06939322
Title: LOG-I - Impact Study of LOG-AFTER Software on Long-term Monitoring of Former Patients (LOG-I - LOG-Impact Study) / Etude d'Impact du Logiciel LOG-AFTER Sur le Suivi à Long Terme Des Anciens Patients (LOG-I - LOG-Impact Study)
Brief Title: LOG-I - Impact Study of LOG-AFTER Software on Long-term Monitoring of Former Patients (LOG-I - LOG-Impact Study)
Acronym: LOG-I
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 49RC25_0035; 2025-A00237-42 (Other: ANSM)
Record Dates: First submitted 2025-03-06; First posted 2025-04-22 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Pediatric Cancer; Cancer Survivor; Hemato-oncologic Patients
Keywords: pediatry; oncology; hematology; radiotherapy; survivorship; preventive care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomization WITH vs WITHOUT use of the software LOG-AFTER designed for survivorship
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Use of the software Log-AFTER (Experimental): Patients are monitored with the help of LOG-AFTER software. Patients are advised to report the completion of the examinations (date and overall conclusion), which allows the software to function properly. The GP is also advised to report any consultations his patient has had with him and to update the date of the examinations if his patient has not done so.
  Interventions: Other: Use of the Log-AFTER software
- WITHOUT Log-After (No Intervention): Patients are monitored without the LOG-AFTER software.

INTERVENTIONS:
Other: Use of the Log-AFTER software — The LOG-AFTER software is used for long-term follow-up care after cancer to empower patients
  Arms: Use of the software Log-AFTER

SUMMARY:
Childhood cancer survivors represent a high-risk population that requires risk-based follow-up. Follow-up recommendations have been harmonized. Education and information practices regarding follow-up recommendations should be personalized, to ensure understanding by all survivors, including those with neurocognitive disorders. Individualized follow-up is necessary to detect complications that may increase morbidity and decrease quality of life, or even increase the risk of early mortality.

In France, the LOG-AFTER software was developed in 2017 by university hospital of Angers and Epiconcept (approved health data host). The main differences with the European procedure concern radiotherapy information, the link with the General practitioner (GP), and the possible addition of information and/or access to therapeutic education in a video format. Indeed, there is the possibility of creating an GP account allowing to receive notifications concerning the follow-up of his patient to be scheduled, to have access to his file summary and his personalized follow-up plan, various information and blank prescription models. LOG-I is a study of the impact of the LOG-AFTER software for the "patient/GP" couple on adherence to follow-up recommendations. LOG-I is interested in all former patients with at least 3 recommendations in their personalized follow-up plan, taking into account the specific population of patients cured of a brain tumor.

DETAILED DESCRIPTION:
Recruitment as long-term follow-up consultations progress. After checking the selection criteria, the investigator informs the patient of the study or the parents of the minor child orally and in writing with delivery of the information letter and answers any questions. If the patient, or their parents for minor patients, agrees to participate, the informed consent form is signed in 2 copies by the different parties. The date of the information and the date of signature of the consent are documented in the patient's source file. Following the inclusion of the patient, randomization is carried out (WITH and WITHOUT use of the LOG-AFTER software).

During this visit, for patients randomized in the LOG-AFTER software, an account is created within 5 days following the consultation.

For all patients (randomized with or without access to LOG-AFTER) the following data are collected in LOG-AFTER:

* Health data: type of first cancer, start and end dates of treatment
* Patient data required for research: gender, month and year of birth, after-effects, psychosocial data (level of education, life as a couple and children if concerned, profession if concerned).

The module to help create the Personalized After-Cancer Plan (PPAC) can be used for everyone and the PPAC is recorded in LOG-AFTER.

The PAM-13 questionnary is completed by the patient.

Contact with the GP : Following the patient's inclusion and randomization in the "WITH access to LOG-after" group, his GP is informed by mail and telephone call. He receives his codes by email via the software.

Patient follow-up : It is organized according to the habits of the specialist and/or his general practitioner.

For patients randomized with access to LOG-AFTER, patients are advised to report the completion of the examinations (date and overall conclusion of the examination), which allows the software to function properly. The GP is also advised to report any consultations his patient has had with him and to update the date of the examinations if his patient has not done so.

Visit at 36 months (+/- 3 months) • For patients randomized to the "LOG-AFTER" group: The patient is contacted 3 years after inclusion by the clinical research associate or reviewed in consultation by the doctor. The follow-up data according to the PPAC are updated if necessary in LOG-AFTER. If necessary, the PPAC can be updated and modified.

The satisfaction questionnaries (Software and Care Pathway) are given (paper format or via the software) to patients and GP. The PAM-13 questionnary is completed again by the patient. A telephone call (doctor or research associate) is made 2 weeks later if not completed with a proposal to do it by telephone.

• For patients randomized to the "usual care" group: The patient is contacted 3 years after inclusion by the clinical research associate or reviewed in consultation by the doctor. The follow-up data according to the PPAC are collected in LOG-AFTER. A satisfaction questionnary on the care pathway (paper format or via software) is sent to patients and GP. The PAM-13 questionnaire is completed again by the patient. A telephone call (doctor or research associate) is made 2 weeks later if not completed with a proposal to do it by telephone.

At the end, an account is created for the patient/GP couple if the patient wishes.

ELIGIBILITY:
Inclusion Criteria:

* Previously treated for cancer or malignant hematological pathology before the age of 25
* Without residual disease or with a stable disease without treatment for 5 years or more
* Owning a computer, smartphone or equivalent I-Pad/tablet with internet access
* Having signed the consent (or their parents if the patient is a minor, or a third party if necessary)
* Having 3 or more recommended screenings in their survivorship care plan
* No access created to LOG-AFTER before the study or having never connected after opening their account if opening an account dating back 24 months or more at the time of inclusion

Exclusion Criteria:

* Patient who has relapsed or developed a second cancer with a post-treatment delay < 5 years
* Patient not covered by a health insurance
* Patient subject to a legal protection measure, patient deprived of liberty by judicial or administrative decision, patient subject to psychiatric care under duress

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2026-11-06 (Estimated); Study Completion 2030-06-06 (Estimated)

PRIMARY OUTCOMES:
PPAC adherence | 3 years
  Evaluate the impact of LOG-AFTER on former patients' adherence to the Personalized After-Cancer Plan (PPAC) for those with at least 3 follow-up examinations.
  (Adherence = For a number of screens between three and six (3-6), adherence is considered adequate if all screens or all but one screen have been completed. For seven or more screens (>7), it is considered adequate if all screens or all but two screens have been completed)

SECONDARY OUTCOMES:
PPAC adherence for survivors of brain tumor treated, at least, with radiotherapy | 3 years
  Evaluate the impact of LOG-AFTER on the adherence of former brain tumor patients who received radiotherapy to the Personalized After-Cancer Plan (PPAC) for those with at least 3 follow-up examinations. (Adherence = For a number of screens between three and six (3-6), adherence is considered adequate if all screens or all but one screen have been completed. For seven or more screens (>7), it is considered adequate if all screens or all but two screens have been completed)
Health status | 3 years
  Establish a descriptive overview of the health status of former patients based on the treatment received =>Descriptive analysis of complications classified by Common Terminology Criteria for Adverse Events (CTCAE) score, including fatigue and cognitive impairment.
  The CTCAE is divided into 5 grades (from grade 1 = Mild; asymptomatic or mild symptoms; diagnosed by clinical examination only; not requiring treatment; to grade 5 = Death related to the adverse event.
PPAC adherence for new cancer survivors partients starting long term follow-up | 3 years
  Describe the impact of LOG-AFTER on the adherence of new cancer survivors starting long term follow-up (Adherence = For a number of screens between three and six (3-6), adherence is considered adequate if all screens or all but one screen have been completed. For seven or more screens (>7), it is considered adequate if all screens or all but two screens have been completed)
PPAC adherence for cancer survivors already involved in long term follow-up before the study | 3 years
  Describe the impact of LOG-AFTER on the adherence of cancer survivors who are not new in long term follow-up (Adherence = For a number of screens between three and six (3-6), adherence is considered adequate if all screens or all but one screen have been completed. For seven or more screens (>7), it is considered adequate if all screens or all but two screens have been completed)
Describe the patient satisfaction | 3 years
  1. satisfaction score from the questionnaire derived from u-MARS for patients randomised with LOG-AFTER.
  2. overall subjective score between 1 and 5 for patients randomised with LOG-AFTER.
  3. qualitative aspect - open field questions, comments
  4. qualitative aspect concerning the care pathway
GP satisfaction | 3 years
  Satisfaction via questionnary derived from of the MARS (Mobile Application Rating Scale) (professionals) for those with access to LOG-AFTER.
  Overall subjective score between 1 (not satified) and 5 (completely satisfied) for those with access to LOG-AFTER.
  Qualitative aspect (free field)
Describe the use | 3 years
  1. number of connections per user
  2. number of connections per of account closures
  3. number of inactive accounts (no use during 6 months or more)
Empowerment | 3 years
  Patient Activation Measure® (PAM®)-13. The score can be 0 (patient not activated) to 100 (patient activated)

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte DEMOOR-GOLDSCHMIDT, Dr, Principal Investigator — University Hospital of Angers
Locations (1):
- University Hospital of Angers, Angers, Maine Et Loire, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://ressources-aura.fr/wp-content/uploads/2023/06/3_Pediatrie-AJA_DEMOOR.pdf